CLINICAL TRIAL: NCT06198738
Title: Correlation Between Silicone-oil Related Ocular Complications and ITMES Score (CLIN-ITEMS)
Acronym: CLIN-ITEMS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cliniche Humanitas Gavazzeni (Other)
Responsible Party: Principal Investigator, Mario R Romano, Professor, Cliniche Humanitas Gavazzeni
Other Study IDs: 344/23
Record Dates: First submitted 2023-12-27; First posted 2024-01-10 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Emulsification of Silicone Oil in Eye Following Surgical Procedure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective, multicentric, observational study aimed to evaluate the correlation between the value of the InTraocular EMulsion of Silicone oil (ITMES) score assessed at clinical examination and silicone oil-related ocular complications. This will allow to clinically validate the ITEMS score, as clinical tool.

Demographic data and clinical findings, including the ITEMS score, of patients undergoing to vitrectomy and silicone oil tamponade or removal of silicone oil or having one silicone oil-filled eye, will be collected at the baseline and at each follow-up visit (at 1-day, 1-, 3- and 6-month after surgery).

The prognostic performance of the ITEMS score will be evaluated in agreement with the TRIPOD statement.

ELIGIBILITY:
Inclusion Criteria: One eye requiring pars plana vitrectomy and silicone oil/heavy silicone oil tamponade, OR pars plana vitrectomy and removal of silicone oil/heavy silicone oil OR one silicone-oil filled eye.

Exclusion Criteria:

* untreated or uncontrolled ocular disease leading to unacceptable higher risk of intra- and post-operative complications, such as uncontrolled ocular inflammation or infection, untreated ocular malignancy and uncontrolled glaucoma;
* uncontrolled severe systemic disease related to significantly higher operative risk;
* pregnant women due to the specific risks related to supine position during surgery, operative time, risks of retrobulbar anesthesia, and intraoperative and postoperative drugs;
* inability to give written consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients meeting the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 323 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Correlation between the value of the ITMES score and any silicone oil-related ocular complication | Baseline, 1 day, 1 month, 3 months and 6 months
  The InTraocular EMulsion of Silicone oil (ITEMS) grading system has been proposed for the assessment of silicone oil emulsion to more reliably quantify the presence and extent of any SO emulsion, applicable in a daily clinical setting and validated through an expert panel consensus procedure (Romano MR, et al, INTRAOCULAR EMULSION OF SILICONE OIL (ITEMS) GRADING SYSTEM: An Evidence-Based Expert-Led Consensus. Retina 2023 Aug 1;43(8):1370-1376)

SECONDARY OUTCOMES:
Correlation between the value of the ITMES score and any single types of intraoperative silicone oil-related ocular complication | Baseline, 1 day, 1 month, 3 months and 6 months
  The InTraocular EMulsion of Silicone oil (ITEMS) grading system has been proposed for the assessment of silicone oil emulsion to more reliably quantify the presence and extent of any SO emulsion, applicable in a daily clinical setting and validated through an expert panel consensus procedure (Romano MR, et al, INTRAOCULAR EMULSION OF SILICONE OIL (ITEMS) GRADING SYSTEM: An Evidence-Based Expert-Led Consensus. Retina 2023 Aug 1;43(8):1370-1376)
Correlation between the value of the ITMES score and any single types of postoperative silicone oil-related ocular complication | Baseline, 1 day, 1 month, 3 months and 6 months
  The InTraocular EMulsion of Silicone oil (ITEMS) grading system has been proposed for the assessment of silicone oil emulsion to more reliably quantify the presence and extent of any SO emulsion, applicable in a daily clinical setting and validated through an expert panel consensus procedure (Romano MR, et al, INTRAOCULAR EMULSION OF SILICONE OIL (ITEMS) GRADING SYSTEM: An Evidence-Based Expert-Led Consensus. Retina 2023 Aug 1;43(8):1370-1376)
Correlation between the value of the ITMES score and postoperative retinal attachment | Baseline, 1 day, 1 month, 3 months and 6 months
  The InTraocular EMulsion of Silicone oil (ITEMS) grading system has been proposed for the assessment of silicone oil emulsion to more reliably quantify the presence and extent of any SO emulsion, applicable in a daily clinical setting and validated through an expert panel consensus procedure (Romano MR, et al, INTRAOCULAR EMULSION OF SILICONE OIL (ITEMS) GRADING SYSTEM: An Evidence-Based Expert-Led Consensus. Retina 2023 Aug 1;43(8):1370-1376)
Correlation between the value of the ITMES score and postoperative best-corrected visual acuity | Baseline, 1 day, 1 month, 3 months and 6 months
  The InTraocular EMulsion of Silicone oil (ITEMS) grading system has been proposed for the assessment of silicone oil emulsion to more reliably quantify the presence and extent of any SO emulsion, applicable in a daily clinical setting and validated through an expert panel consensus procedure (Romano MR, et al, INTRAOCULAR EMULSION OF SILICONE OIL (ITEMS) GRADING SYSTEM: An Evidence-Based Expert-Led Consensus. Retina 2023 Aug 1;43(8):1370-1376)